CLINICAL TRIAL: NCT04068597
Title: An Open-label Phase I/IIa Study to Evaluate the Safety and Efficacy of CCS1477 as Monotherapy and in Combination in Patients With Advanced Haematological Malignancies.
Brief Title: Study to Evaluate CCS1477 (Inobrodib) in Haematological Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CellCentric Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CCS1477-02
Record Dates: First submitted 2019-08-12; First posted 2019-08-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Haematological Malignancy; Acute Myeloid Leukemia; Non Hodgkin Lymphoma; Multiple Myeloma; Higher-risk Myelodysplastic Syndrome; Peripheral T Cell Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, T-Cell, Peripheral | interventions — CCS1477; pomalidomide; Dexamethasone; Azacitidine; venetoclax; Bortezomib; ixazomib; Lenalidomide; daratumumab

STUDY DESIGN:
Intervention Model Description: The RP2D/MTD dose will be determined in Parts A and B. Parts C, D, E and F of the study may recruit patients concurrently.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- CCS1477 dose escalation NHL/MM (Experimental): CCS1477 monotherapy
  Interventions: Drug: CCS1477
- CCS1477 dose escalation AML/Higher risk MDS (Experimental): CCS1477 monotherapy
  Interventions: Drug: CCS1477
- CCS1477 monotherapy expansion and combination dose finding and expansion NHL (Experimental): CCS1477 monotherapy, CCS1477 combination with lenalidomide
  Interventions: Drug: CCS1477; Drug: Lenalidomide
- CCS1477 monotherapy expansion and combination dose finding and expansion - MM (Experimental): CCS1477 monotherapy, CCS1477 combination with pomalidomide-dexamethasone, CCS1477 combination with bortezomib-dexamethasone, CCS1477 combination with ixazomib-dexamethasone, CCS1477 combination with elranatamab, CCS1477 combination with teclistamab, CCS1477 combination with lenalidomide, CCS1477 combination with lenalidomide and daratumumab
  Interventions: Drug: CCS1477; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib; Drug: Ixazomib; Drug: Elranatamab; Drug: Teclistamab; Drug: Lenalidomide; Drug: Daratumumab
- CCS1477 monotherapy expansion and combination dose finding and expansion - AML (Experimental): CCS1477 monotherapy, CCS1477 combination with azacitidine, CCS1477 combination with azacitidine and venetoclax
  Interventions: Drug: CCS1477; Drug: Azacitidine; Drug: Venetoclax
- CCS1477 monotherapy expansion and combination dose finding and expansion - Higher risk MDS (Experimental): CCS1477 monotherapy, CCS1477 combination with azacitidine
  Interventions: Drug: CCS1477; Drug: Azacitidine

INTERVENTIONS:
Drug: CCS1477 — Oral capsule
Drug: Pomalidomide — oral capsule
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Dexamethasone — oral tablet
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Azacitidine — Powder suspension for Injection
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - AML; CCS1477 monotherapy expansion and combination dose finding and expansion - Higher risk MDS
Drug: Venetoclax — Oral tablet
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - AML
Drug: Bortezomib — Powder for solution for injection
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Ixazomib — Oral capsule
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Elranatamab — Solution for injection
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Teclistamab — Solution for injection
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM
Drug: Lenalidomide — Oral capsule
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM; CCS1477 monotherapy expansion and combination dose finding and expansion NHL
Drug: Daratumumab — Solution for injection, concentrate for solution for infusion
  Arms: CCS1477 monotherapy expansion and combination dose finding and expansion - MM

SUMMARY:
A Phase 1/2a study to assess the safety, tolerability, PK and biological activity of CCS1477 (inobrodib) in patients with Non-Hodgkin Lymphoma, Multiple Myeloma, Acute Myeloid Leukaemia or High Risk Myelodysplastic syndrome.

DETAILED DESCRIPTION:
This includes patients with Peripheral T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Provision of consent
* ECOG performance status 0-2
* Patients with confirmed (per standard disease specific diagnostic criteria), relapsed or refractory haematological malignancies (NHL, MM and AML)
* Must have previously received standard therapy
* Adequate organ function

Exclusion Criteria:

* Intervention with any chemotherapy, investigational agents or other anti-cancer drugs within 14 days or 5 half-lives of the first dose
* Major surgical procedure or significant traumatic injury within 4 weeks of the first dose of study treatment
* Strong inhibitors of CYP3A4 or CYP3A4 substrates with a narrow therapeutic range taken within 2 weeks of the first dose of study treatment
* Strong inducers of CYP3A4 within 4 weeks of the first dose of study treatment
* Patients should discontinue statins prior to starting study treatment
* CYP2C8 substrates with a narrow therapeutic range taken within 2 weeks of the first dose of study treatment
* Any unresolved reversible toxicities from prior therapy >CTCAE grade 1 at the time of starting study treatment (except alopecia and grade 2 neuropathy)
* Any evidence of severe or uncontrolled systemic diseases
* Any known uncontrolled inter-current illness
* QTcF prolongation (> 470 msec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-08-09 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | Up to 12 months
  Treatment-related adverse events and serious adverse events
Incidence of laboratory abnormalities | Up to 12 months
  Laboratory abnormalities characterised by type, frequency, severity and timing

SECONDARY OUTCOMES:
Response rate | Up to 12 months
  Defined as number of patients who have a response according to
  * RECIL criteria (NHL)
  * IMWG criteria (Multiple myeloma)
  * ELN recommendations 2017 (AML)
Duration of Response | Up to 12 months
  Defined as the time from start of treatment until disease progression
AUC of CCS1477 | 35 days
  Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last measurable concentration of CCS1477
Cmax of CCS1477 | 35 days
  Maximum observed plasma concentration (Cmax) of CCS1477

CONTACTS AND LOCATIONS:
Overall Officials: Tim Somervaille, Principal Investigator — The Christie NHS Foundation Trust
Locations (39):
- United States (6):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Community Health Network, Indianapolis, Indiana
  - The Center for Cancer and Blood Disorders (CCBD), Bethesda, Maryland
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Penn Medicine - Abramson Cancer Center Perelman, Philadelphia, Pennsylvania
- France (2):
  - Institute Bergonie, Bordeaux
  - Gustave Roussy, Villejuif
- Spain (12):
  - Hospital Germans Trias i Pujol/ ICO Badalona, Badalona
  - University Hospital Vall D'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - ICO L'Hospitalet (Instituto Catalán de Oncología), Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Universidad de Navarra, Pamplona
  - Hospital Universitario y Politécnico La Fe de la Comunidad Valenciana, Valencia
- Karolinska Comprehensive Cancer Center, Stockholm, Sweden
- United Kingdom (18):
  - The Royal Marsden, Sutton, Surrey
  - The Clatterbridge Cancer Centre NHS Foundation Trust,, Bebington
  - University Hospitals Bristol, Bristol
  - University Hospital of Wales, Cardiff
  - Royal Derby Hospital, Derby
  - Western General Hospital, Edinburgh
  - Gartnavel General Hospital, Glasgow
  - Leicester Royal Infirmary, Leicester
  - St Bartholomew's Hospital, London
  - Sarah Cannon Research Institute UK, London
  - NIHR University College London Clinical Research Facility, London
  - Imperial College, London
  - The Christie Hospital, Manchester
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Cancer and Haematology Centre, Oxford
  - University Hospital of Southampton, Southampton
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
At this stage, is not currently planned that any IPD information will be shared with other researchers outside of the Sponsor and Clinical Research Organisations involved in the conduct of this study.